CLINICAL TRIAL: NCT04204239
Title: A Review of Test Procedures From Different Health Care Professions With Regard to Their Suitability for the Early Detection of Cognitive Impairments in Persons Aged 60 and Older: A Validation Study
Brief Title: Validation Study SCOBES-AR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FH Joanneum Gesellschaft mbH (Industry)
Collaborators: Austrian Research Promotion Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: Validation study SCOBES-AR
Record Dates: First submitted 2019-12-11; First posted 2019-12-18 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Decline; Cognitive Deficit; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose of the study The purpose of this study is to evaluate five tests to see if they are suitable for the early detection of cognitive impairment in people over the age of 60. These test procedures record the movement pattern and gait pattern, the reaction time, so-called instrumental activities of daily life (e.g. shopping or preparing meals), nutritional behaviour and the relevant sense of smell. The results are compared with those of a diagnostic procedure already in use.

DETAILED DESCRIPTION:
Improved living conditions and health care are making people in Austria older and older. However, OECD data show that this happens with a lower quality of life compared to other EU member states. One factor influencing the quality of life is individual functionality at the physical and cognitive levels. Physical functionality is obvious, but cognitive impairment is preceded by a long latency phase in which subtle limitations of executive functions exist. Studies have shown that early detection of dementia through screening and early intervention can make an important contribution to a favourable course of treatment. Measures of early detection and prevention for the prevention of clinical occurrence thus move into focus. Current clinical diagnostic procedures such as cerebrospinal fluid diagnostics and MRI are not suitable for population-based early detection. Augmented Reality (AR) techniques represent an innovative basis for the development of information and communication technology (ICT) based assessment procedures. Real objects are extended by means of smartphones with virtual objects and tasks as test objects of screening. Parallel measurements of multiple parameters, automatic action recording and semi-automated evaluations provide detailed results.

The project SCOBES-AR (Smart Cognition & Behaviour Screening powered by Augmented Reality) is funded by the Austrian Research Promotion Agency (FFG) and has a maximum duration of five years (September 2023). Through the cooperation of various health science and technical study programmes (dietology, occupational therapy, health and nursing, health management in tourism/sports science laboratory, information management, speech therapy, physiotherapy) of FH JOANNEUM, a screening instrument for the early detection of neurocognitive deficits is to be developed. The aim is to establish a multimodal tool for sustainable use in the health care system. The project thus takes up the impact goals of the Austrian dementia strategy and aims to develop a multimodal screening instrument for the early detection of functional impairments (on a cognitive and physical level) in middle and old age for outpatient care. In Phase I of the project, the evidence base for a valid instrument will be developed - The focus is on assessment selection, data protection and implementation in an AR environment. The evaluation and validation of the prototype and the AR environment are carried out in phase I and phase II respectively. In Phase III, a business model for sustainable use in the health care system with possibilities in the big data area will be developed for the finalized instrument. The present study protocol only describes the validation study in phase I of the project.

• Research objectives in phase I of the project In order to realize the main goal of the project, to develop a multimodal and low-threshold screening instrument embedded in an AR environment for the early detection of functional limitations on cognitive for outpatient care, comprehensive preliminary investigations are necessary.

The validation study presented here is one of these preliminary investigations. Five test procedures are to be tested to determine whether they are suitable for the early detection of cognitive impairments in people aged 60 and over and thus whether the evidence base for a valid instrument can be established. Different functionalities such as movement pattern & gait pattern, reaction time, instrumental activities of daily life (iADL) will be recorded and evaluated. Examples of iADLs are shopping, financial regulation, mobility or preparing meals. Nutritional behaviour is also evaluated, since, for example, adherence to a Mediterranean diet is associated with a lower risk of various age-related diseases, including dementia. Another possible predictive factor for the development of neurocognitive impairment is the decrease in olfactory performance, which is why olfactory performance is also measured. The collected data should be compared with the established test battery "Cognitive Functions Dementia" (CFD), which is widely used in neuropsychological practice, to clarify cognitive impairments and thus be validated. The combination of the collected data results in a comprehensive functional status picture of the tested persons. Due to the extensive test setting with different test items, SCOBES-AR offers a comprehensive view of the cognitive and physical functionalities of the test person. It allows the Focus on existing reserves and capacities of the test person and not on their deficits.

The results of the present validation study will be used at the end of the project to collect the above-mentioned - or similar - functionalities via assessments, which are partly implemented in an Augmented Reality environment.

* Primary hypothesis of the study The planned tests are suitable for the early detection of cognitive impairment in people over 60 years of age.
* Secondary hypotheses of the study The primary target group (people aged 60 and over) is interested in recognising functional (cognitive and physical) limitations at an early stage in order to be able to work specifically on improving them.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 60-75 years
* Interested in participating in the study
* Signing a written informed consent form

Exclusion Criteria:

* Persons who are not legally competent (Austrian adult protection law)
* Clinical diagnosis of dementia or MCI (Mild Cognitive Impairment)
* Clinical diagnosis of mental illness (e.g. depression or psychosis)
* Reduced mobility (sidekick, wheelchair)
* No compensation for visual or hearing impairment
* Insufficient knowledge of German

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the city of Graz and Graz suburbs
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Erlangen Test of Activities of daily living in Persons with Mild Dementia or Mild Cognitive impairment (ETAM) | By completing the entire test set, an average of 2 hours
  For three Items the performance is evaluated on a seven-level scale (0-6 points). The execution of an item is subdivided into six sub-steps so that the test persons receive one point for each error-free sub-step. A four-step scale (0-3 points) was used for two items with a less complex structure (alarm clock and tea). The total value ranges from 0-30 points.
Brief Smell Identification Test (B-SIT) | By completing the entire test set, an average of 2 hours
  The test person should recognize 12 different odorous substances and choose from a four-step multiple-choice question. A total odour score results from the number of correctly identified odours, whereby higher values stand for a better odour performance (>9 recognised odours).
Reaction test (TDS) | By completing the entire test set, an average of 2 hours
  Eye to hand reaction, eye to leg reaction, complex reaction capability; the time required (seconds/milliseconds) for the completion is recorded.
Dual-Task-Assessment (DTA) | By completing the entire test set, an average of 2 hours
  Measures the influence of a cognitive task on the gait pattern. Impaired subjects show a stronger change of different gait parameters. The gait speed, cadence, stride length, stride variance and gait phases are measured.
Mediterranean Diet Adherence Score (MEDAS) | By completing the entire test set, an average of 2 hours
  14-Elements-Screeningtool for the evaluation of the adherence to the Mediterranean diet. The maximum score is 14 points and indicates full compliance with the Mediterranean diet.

SECONDARY OUTCOMES:
Cognitive Functions Dementia (CFD) | By completing the entire test set, an average of 2 hours
  A digital test set for the early diagnosis of dementia. It contains tests for verbal learning and memory skill, working memory, measurement of attention, cognitive flexibility, information processing speed, visuoconstruction, object naming and verbal fluency.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Staubmann, BSc MSc, Study Director — University of Applied Sciences, FH JOANNEUM
Locations (1):
- University of Applied Sciences, FH JOANNEUM, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hebestreit K, Yahiaoui-Doktor M, Engel C, Vetter W, Siniatchkin M, Erickson N, Halle M, Kiechle M, Bischoff SC. Validation of the German version of the Mediterranean Diet Adherence Screener (MEDAS) questionnaire. BMC Cancer. 2017 May 18;17(1):341. doi: 10.1186/s12885-017-3337-y. PMID 28521737
- [Background] American Occupational Therapy Association (Hrsg.). (2018). Das Framework der AOTA. Gegenstandsbereich, Prozesse und Kontexte in der ergotherapeutischen Praxis. Bern: Hogrefe.
- [Background] Doty RL, Marcus A, Lee WW. Development of the 12-item Cross-Cultural Smell Identification Test (CC-SIT). Laryngoscope. 1996 Mar;106(3 Pt 1):353-6. doi: 10.1097/00005537-199603000-00021. PMID 8614203
- [Background] Hendry K, Quinn TJ, Evans JJ, Stott DJ. Informant single screening questions for delirium and dementia in acute care--a cross-sectional test accuracy pilot study. BMC Geriatr. 2015 Feb 25;15:17. doi: 10.1186/s12877-015-0016-1. PMID 25885022
- [Background] Hunter SW, Divine A, Frengopoulos C, Montero Odasso M. A framework for secondary cognitive and motor tasks in dual-task gait testing in people with mild cognitive impairment. BMC Geriatr. 2018 Sep 3;18(1):202. doi: 10.1186/s12877-018-0894-0. PMID 30176796
- [Background] Jahn, T. & Heßler, J. B. (2017). Handanweisung Kognitive Funktionen Demenz (Kurzbezeichung CFD). Mödling: Schufried GmbH
- [Background] Juraszovich, B.; Sax, G.; Rappold, E.; Pfabigan, D. & Stewig, F. (Hg). (2015). Demenzstrategie Gut Leben mit Demenz. Wien: Bundesministerium für Gesundheit und Sozialministerium; 2015.
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Background] Lin KC, Wu YF, Chen IC, Tsai PL, Wu CY, Chen CL. Dual-task performance involving hand dexterity and cognitive tasks and daily functioning in people with schizophrenia: a pilot study. Am J Occup Ther. 2015 May-Jun;69(3):6903250020p1-7. doi: 10.5014/ajot.2014.014738. PMID 25871598
- [Background] Luttenberger K, Reppermund S, Schmiedeberg-Sohn A, Book S, Graessel E. Validation of the Erlangen Test of Activities of Daily Living in Persons with Mild Dementia or Mild Cognitive Impairment (ETAM). BMC Geriatr. 2016 May 26;16:111. doi: 10.1186/s12877-016-0271-9. PMID 27229937
- [Background] Lourida I, Soni M, Thompson-Coon J, Purandare N, Lang IA, Ukoumunne OC, Llewellyn DJ. Mediterranean diet, cognitive function, and dementia: a systematic review. Epidemiology. 2013 Jul;24(4):479-89. doi: 10.1097/EDE.0b013e3182944410. PMID 23680940
- [Background] Yahiaoui-Doktor M, Luck T, Riedel-Heller SG, Loeffler M, Wirkner K, Engel C. Olfactory function is associated with cognitive performance: results from the population-based LIFE-Adult-Study. Alzheimers Res Ther. 2019 May 10;11(1):43. doi: 10.1186/s13195-019-0494-z. PMID 31077241
- See also: OECD. Health at a Glance 2017: OECD Indicators, OECD Publishing, 2017, Paris. — https://www.oecd-ilibrary.org/sites/health_glance-2017-en/index.html?itemId=/content/publication/health_glance-2017-en